CLINICAL TRIAL: NCT06688162
Title: Minimally Invasive Soft Channel Brain Haemorrhage Evacuation for Acute Basal Ganglia Haemorrhage--Small Hemorrhage Evacuation (MIRACLE-S)
Acronym: MIRACLE-S
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Fudan University (Other); Linyi People's Hospital (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, President, Head of Neurology, Principal Investigator, Clinical Professor, Xuanwu Hospital of Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIRACLE-S
Record Dates: First submitted 2024-10-17; First posted 2024-11-14 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Placebo Comparator): Usual Care
  Interventions: Other: Usual Care
- Minimally Invasive Soft Channel Brain Haemorrhage Evacuation (scMIS) (Experimental): Minimally Invasive Soft Channel Brain Haemorrhage Evacuation(scMIS)
  Interventions: Procedure: Minimally Invasive Soft Channel Brain Haemorrhage Evacuation (scMIS)

INTERVENTIONS:
Other: Usual Care — During the study treatment and follow-up periods, patients are to receive usual standard of care according to published guidelines for acute stroke care. It is anticipated that background care may include the use of other treatments including drugs and interventions.
  Arms: Usual Care
Procedure: Minimally Invasive Soft Channel Brain Haemorrhage Evacuation (scMIS) — This technique is based on the study of hematoma anatomy, cerebral vascular anatomy, and neural fiber structure anatomy in basal ganglia hemorrhage to determine the optimal surgical (catheter insertion) path. By applying stereogeometric principles, it allows for simple yet precise localization. Through surgical steps including puncture, aspiration, liquefaction (intermittent infusion of urokinase or alteplase), and external drainage, the hematoma can be completely removed in stages over a short period. This ensures that hematoma clearance and decompression of the brain occur simultaneously, achieving a minimally invasive intracerebral hemorrhage evacuation technique with a gradual reduction in intracranial pressure.
  Arms: Minimally Invasive Soft Channel Brain Haemorrhage Evacuation (scMIS)

SUMMARY:
The objective of this study is to determine whether minimally invasive soft channel brain hemorrhage evacuation (scMIS), compared to usual care, leads to superior functional recovery as measured by utility-weighted modified Rankin Scale (UW-mRS) scores at 6 months in patients with basal ganglia intracerebral hemorrhage (ICH) of 20 ≤ volume ≤ 30 ml.

ELIGIBILITY:
* Inclusion Criteria:

  1. Adults (18 - 80 years) ;
  2. The clinical diagnosis is acute intracerebral hemorrhage, confirmed by imaging;
  3. Onset within 48 hours, and surgery can be initiated within 48 hours;
  4. Basal ganglia hemorrhage, with a bleeding volume of 20 ≤ volume ≤ 30 ml;
  5. Reduced level of consciousness (GCS 9-14);
  6. Pre-stroke mRS score≤1 points;
  7. Systolic blood pressure <140 mmHg before randomisation;
  8. Informed consent obtain accordingly to local regulations.
* Exclusion Criteria:

  1. Definite evidence the ICH is secondary to a structural abnormality in the brain (eg arteriovenous malformation, intracranial aneurysm, tumour, trauma, cerebral venous thrombosis) or previous thrombolysis or neurointerventional surgery.
  2. A high likelihood that the patient will not adhere to the study treatment and follow-up regimen.
  3. Platelet count < 100,000, INR > 1.4.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional recovery according to UW-mRS assessed at 6 months | 6 months
  Utility weighted modified rankin scale scores is to map functional status (modified Rankin Scale [mRS] scores) and health-related quality of life on the European Quality of Life 5-dimensional questionnaire (EQ-5D) to derive utility-weighted (UW) stroke outcome measures.

SECONDARY OUTCOMES:
Discharge at Day 7 (yes vs. no) | 7 days after randomization
  Discharge status will be assessed at Day 7
Total length of intensive care unit stay. | During hospitalisation up to 6 months after randomization
  The complete length of time a patient is admitted to the intensive care unit (ICU)
Ordinal analysis of modified Rankin Scale [mRS] scores at 28 days | 28 days after randomization
  Ordinal analysis of modified Rankin Scale [mRS] score:
  0 =No symptoms at all.1 =No significant disability despite symptoms, able to carry out all usual duties and activities.2 =Slight disability, unable to carry out all previous activities but able to look after own affairs without assistance.3 =Moderate disability requiring some help, but able to walk without Assistance.
  4 =Moderate severe disability, unable to walk without assistance and unable to attend to own bodily needs without assistance.5 =Severe disability, bedridden incontinent, and requiring constant nursing care and attention.6 =Dead.
The following at 6-months: ordinal analysis of modified Rankin Scale [mRS] scores 3-6 | 6-months after randomization
  Proportion of subjects with modified Rankin Scale [mRS] 3-6 at 6 months after randomization
The following at 6-months: ordinal analysis of modified Rankin Scale [mRS] scores 3-5 | 6-months after randomization
  Proportion of subjects with modified Rankin Scale [mRS] 3-5 at 6 months after randomization
The following at 6-months: ordinal analysis of modified Rankin Scale [mRS] scores 0-6 | 6-months after randomization
  Modified Rankin Scale [mRS] score at 6 months analysed as an ordinal outcome (categories 0 to 6).
The following at 6-months: AMC Linear Disability Score(ALDs) | 6-months after randomization
  The AMC (Academic Medical Center) Linear Disability Score (ALDs) is a calibrated generic item bank designed to measure physical disability levels in patients. The ALDs is a sensitive and generic scale that encompasses a broader range of activities compared to the Rankin assessment. The key distinction between the ALDs and the Rankin assessment is that the ALDs provides a linear disability score based on patient-reported outcomes, while the Rankin score is an ordinal assessment determined by a rater.
The following at 6-months: EuroQoL Group 5-Dimension self-report questionnaire (EQ-5D) | 6-months after randomization
  An EQ-5D score, also referred to as an EQ-5D value index or utility, quantifies a person's health status on a scale from 1 (full health) to 0 (equivalent to being dead). Negative values may be assigned to health states considered worse than death.The score is calculated using a formula that applies specific weights to each level in the various dimensions of the EQ-5D, with these weights derived from a value set that includes index values for all possible EQ-5D states.
Days of hospitalization | During hospitalisation up to 6 months after randomization
  Length of stay in hospital

OTHER OUTCOMES:
Safety outcomes | Throughout the entire study period up to 6 months after randomization
  Mortality, rebleeding, infections, and other serious adverse events (SAEs) recorded throughout the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: XunMing JI, PhD, Principal Investigator — Capital Medical University
Locations (1):
- Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No